CLINICAL TRIAL: NCT01884402
Title: Observational,Post-authorization Prospective Study to Develop and Validate a Prognostic Tool for Optimizing Therapy in Patients With Hepatitis C Virus (HCV) Genotype 1 and 4.
Brief Title: Observational,Prospective Study to Develop and Validate a Prognostic Tool to Optimize Therapy in Patients With HCV G1/4
Acronym: OPTIM
Status: Completed | Type: Observational
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: FPS-PEG-2010-01
Record Dates: First submitted 2013-06-18; First posted 2013-06-24 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pegasys, injection subcutaneous: HCV patients monoinfected or coinfected genotype 1/4 treated with Peginterferon alfa-2a and Ribavirin
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Peginterferon alfa-2a — Treatment as usual clinical practice
  Other Names: Pegasys
Drug: Ribavirin — Treatment as usual clinical practice
  Other Names: Copegus

SUMMARY:
Primary objective:

• Develop and validate a tool towards patients with chronic hepatitis C genotype 1 and 4 to allow optimize treatment.

DETAILED DESCRIPTION:
This Tool:

1. Predicting the overall impact of prognostic factors (including the new factor of genetic polymorphism of the IL28B) on Sustained Viral Response (SVR).
2. Identify those patients most likely to respond.
3. Therapy and therefore optimize resources

The validation tool will check into clinical practice its predictive power (it will consider its ability to calibrate and discriminate) and make correct inferences and interpretations of the scores obtained when applying.

ELIGIBILITY:
Inclusion Criteria:

* Patients with > 18 years old.
* Patients diagnosed with chronic hepatitis C in the presence of HCV RNA in plasma that meet criteria for initiating antiviral therapy in routine clinical practice conditions.
* Patients Genotype 1 and 4.
* Patients with the results of all the factors evaluable at the time of inclusion.
* Patients who have accepted their participation in the study through informed consent.

Exclusion Criteria:

* Patients previously treated with interferon (IFN) and ribavirin (RBV).
* Patients with genotype 2, 3, 5 and 6.
* Patients with co-infection with hepatitis B.
* Patients with other liver diseases.
* Patients with any contraindications to the drugs used in the treatment of hepatitis C.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis C genotype 1 and 4 mono-or co-infected with HIV who meet the selection criteria described.
Sampling Method: Non-Probability Sample
Enrollment: 770 (Actual)
Dates: Start 2010-10; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Sustained Viral Response (RVS) | 1 ½ years (72 weeks)
  Measurement of HCV RNA negativization 24 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Romero-Gómez, Medicine, Principal Investigator — Hospital de Valme & ciberEHD
Locations (2):
- Spain (2):
  - Fundación Pública Andaluza para la Gestión de la investigación en salud de Sevilla (FISEVI), Seville, Sevilla
  - Fundación Pública Andaluza para la Gestión de la investigación en salud de Sevilla (FISEVI), Seville